CLINICAL TRIAL: NCT03340727
Title: Randomized Controlled Trial of Home Therapy With Caffeine Citrate in Moderately Preterm Infants With Apnea of Prematurity
Brief Title: Moderately Preterm Infants With Caffeine at Home for Apnea (MoCHA) Trial
Acronym: MoCHA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Futility
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NICHD-NRN-0056; UG1HD034216 (NIH); UG1HD027904 (NIH); UG1HD021364 (NIH); UG1HD027853 (NIH); UG1HD040689 (NIH); UG1HD040492 (NIH); UG1HD027851 (NIH); UG1HD087229 (NIH); UG1HD053109 (NIH); UG1HD068278 (NIH); UG1HD068244 (NIH); UG1HD068263 (NIH); UG1HD027880 (NIH); UG1HD053089 (NIH); UG1HD087226 (NIH); U10HD036790 (NIH)
Record Dates: First submitted 2017-11-03; First posted 2017-11-13 (Actual); Results first posted 2024-06-28 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Apnea of Prematurity
Keywords: Moderate preterm infant; Caffeine citrate
MeSH Terms: conditions — Apnea | interventions — caffeine citrate

STUDY DESIGN:
Intervention Model Description: Sample size for this trial will be flexible: the trial will be stopped for efficacy or futility based on pre-determined statistical thresholds or based on study drug availability.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Caffeine Citrate (Experimental): Caffeine citrate at 10 mg/kg/dose (5 mg/kg caffeine base) daily, in hospital. Infants will continue at home on the same dose of caffeine citrate for the first 28 days after hospital discharge.
  Interventions: Drug: Caffeine Citrate
- Placebo (Placebo Comparator): Placebo contains all of the excipients except for the active ingredient, caffeine citrate, (a volume equivalent to 10 mg/kg of caffeine citrate) and given daily. Infants will be continued at home on the same dose of placebo for the first 28 days after hospital discharge.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Caffeine Citrate — The study intervention is caffeine citrate given once daily at 10 mg/kg/day. It is given orally, before hospital discharge and 28 days after discharge.
  Arms: Caffeine Citrate
Drug: Placebo — The study intervention is placebo given once daily at a volume equivalent to 10 mg/kg of caffeine citrate. It is given orally, before hospital discharge and 28 days after discharge.
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the effect of continuing treatment with caffeine citrate in the hospital and at home in moderately preterm infants with resolved apnea of prematurity on days of hospitalization after randomization.

DETAILED DESCRIPTION:
Study subjects will be patients in the NICU at one of the participating hospitals at a Neonatal Research Network site. Infants who meet the eligibility criteria will be randomized to either caffeine citrate at 10 mg/kg/dose or placebo (equal volume of all the excipients except for the active ingredient, caffeine citrate) to be given daily beginning within 72 hours of open label caffeine discontinuation. The infant may still require hospitalization for observation after discontinuation of open label caffeine or for other discharge issues such as temperature control or feeding tolerance.

Once deemed ready for discharge, infants will be continued at home on the same dose of caffeine citrate or placebo for the first 28 days after hospital discharge. On the day of discharge, the parent will be supplied with 28 numbered vials with oral caffeine citrate (intervention group) or placebo at an equivalent volume (placebo group).

The parents will be educated by the research nurse, discharge nurse, physician, or pharmacist on storage and administration of study medication. A member of the research team will contact the parents to obtain post-discharge information within 72 hours after discharge, once a week for the first 4 weeks, and biweekly during the weeks 5 to 8 after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Inborn and outborn infants of 29 0/7 to 33 6/7 weeks gestational age at birth
* admitted to hospitals of the NICHD NRN who, are at time of enrollment:
* ≤35 6/7 weeks post-menstrual age at the time of randomization
* Receiving caffeine with plan to discontinue treatment or just discontinued caffeine treatment
* Receiving feeds at a volume of ≥120 ml/kg/day by oral and/or tube feeding
* Ability to start study medication within 72 hours after stopping caffeine

Exclusion Criteria:

* On respiratory therapy (oxygen more than room air equivalent for high altitude sites, nasal cannula, continuous positive pressure ventilation, and/or mechanical ventilation)
* Infants who would otherwise be discharged home on apnea monitor due to underlying disease or family history, including history of a sibling with sudden infant death syndrome
* Parental request for apnea monitor
* Congenital heart disease other than atrial septal defect, ventricular septal defect, or patent ductus arteriosus
* Neuromuscular conditions affecting respiration
* Major congenital malformation and/or genetic disorder
* Plans to transfer to a non-NRN site before discharge
* Unable to obtain parental or guardian consent

Ages: 29 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 827 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Waldemar Carlo, MD, Principal Investigator — University of Alabama at Birmingham
Locations (16):
- United States (16):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - Emory University, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - University of New Mexico, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Per NIH Data Sharing Plan

REFERENCES:
- [Derived] Carlo WA, Eichenwald EC, Carper BA, Bell EF, Keszler M, Patel RM, Sanchez PJ, Goldberg RN, D'Angio CT, Van Meurs KP, Hibbs AM, Ambalavanan N, Cosby SS, Newman NS, Vohr BR, Walsh MC, Das A, Ohls RK, Fuller J, Rysavy MA, Ghavam S, Brion LP, Puopolo KM, Moore R, Baack ML, Colaizy TT, Baserga M, Osman AF, Merhar SL, Poindexter BB, DeMauro SB, Kumar V, Cotten CM; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Extended Caffeine for Apnea in Moderately Preterm Infants: The MoCHA Randomized Clinical Trial. JAMA. 2025 Jun 24;333(24):2154-2163. doi: 10.1001/jama.2025.5791. PMID 40294395

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Infants were recruited into the study based on eligibility and parental/guardian consent. Baseline characteristics of the mother were collected (with consent) for use in statistical analysis.
Groups:
- Caffeine Citrate: Daily weight-adjusted doses of Caffeine Citrate while in the hospital, followed by 4 weeks of at home administration by parent/guardians
- Placebo: Daily weight-adjusted doses of Placebo while in the hospital, followed by 4 weeks of at home administration by parent/guardians
Period: Overall Study
Arm/Group | Caffeine Citrate | Placebo
Started | 416 | 411
Completed In-hospital Stay | 390 | 397
Completed (Completed At-home Portion) | 345 | 351
Not Completed | 71 | 60
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 31 | 35
Not completed — Still in hospital at 48 0/7 wks Post-menstrual Age (PMA) | 1 | 1
Not completed — Transferred to another facility | 10 | 7
Not completed — Withdrawal by Subject | 28 | 17

BASELINE CHARACTERISTICS:
Population: The study recruited infants based on eligibility and parental/guardian consent. Baseline characteristics of the mother were collected (with consent) for use in statistical analysis.
Groups:
- Caffeine: Daily weight-adjusted doses of Caffeine Citrate while in the hospital, followed by 4 weeks of at home administration by parent/guardians
- Total: Total of all reporting groups
Arm/Group | Caffeine | Placebo | Total
Number analyzed (Participants) | 416 | 411 | 827
Age, Continuous [Mean (Standard Deviation); unit: years] — Mother's age at time of birth of infant
  years | 30 (5.8) | 29.9 (5.8) | 29.9 (5.8)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Sex assigned to infant a birth
  Participants
    Female | 213 | 207 | 420
    Male | 203 | 204 | 407
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Self-reported race of Mother
  Participants
    American Indian or Alaskan Native | 7 | 12 | 19
    Asian | 12 | 9 | 21
    Black | 110 | 110 | 220
    More Than One Race | 3 | 2 | 5
    Native Hawaiian or Other Pacific Islander | 4 | 4 | 8
    Unknown | 2 | 2 | 4
    Unknown or Not Reported | 13 | 11 | 24
    White | 265 | 261 | 526
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Self-reported ethnicity of mother
  Participants
    Hispanic or Latino | 63 | 54 | 117
    Not Hispanic or Latino | 338 | 345 | 683
    Unknown | 2 | 2 | 4
    Unknown or Not Reported | 13 | 10 | 23
Marital status [Count of Participants; unit: Participants] — Mother's marital status at time of birth of infant
  Participants
    Married | 213 | 233 | 446
    Single | 200 | 175 | 375
    Unknown | 3 | 3 | 6
Mothers education, Customized [Count of Participants; unit: Participants] — Highest level of education of Mother at time of birth of infant
  Participants
    8th grade or less | 9 | 5 | 14
    9th to 12th grade | 33 | 22 | 55
    College degree | 68 | 75 | 143
    Graduate degree | 38 | 38 | 76
    High School degree | 86 | 102 | 188
    Partial college/Associate degree | 93 | 90 | 183
    Trade or technical school | 10 | 10 | 20
    Unknown | 79 | 69 | 148
Mothers insurance, Customized [Count of Participants; unit: Participants] — Type of insurance of Mother at time of birth of infant
  Participants
    Private | 207 | 213 | 420
    Public | 203 | 190 | 393
    Self-pay/uninsured | 6 | 7 | 13
    Unknown | 0 | 1 | 1
Gravidity [Median (Inter-Quartile Range); unit: years] | 2.5 [1 to 4] | 2 [1 to 4] | 2 [1 to 4]
Parity [Median (Inter-Quartile Range); unit: years] | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3]
Gestational Age [Mean (Standard Deviation); unit: weeks] — Gestational age of infant at time of birth
  weeks | 31.2 (1.2) | 31.2 (1.2) | 31.2 (1.2)
Birth weight of infant [Mean (Standard Deviation); unit: grams] | 1545 (358.1) | 1564.3 (357.4) | 1554.6 (357.7)
Apgar score of Infant at 1 minute after birth [Median (Inter-Quartile Range); unit: score] — Apgar scoring involves evaluating 5 vital signs of newborns: Appearance/color, Pulse/heart rate, Grimace response/reflexes, Activity/muscle tone, and Respiration. Each sign receives a score between 0 and 2, with high score indicating better health. The Total Apgar Score is calculated by summing the individual aspect scores and ranges from 0 to 10, with higher scores indicating better health.
  score | 6 [4 to 8] | 6 [4 to 8] | 6 [4 to 8]
Apgar score of Infant at 5 minutes after birth [Median (Inter-Quartile Range); unit: score] — Apgar scoring involves evaluating 5 vital signs of newborns: Appearance/color, Pulse/heart rate, Grimace response/reflexes, Activity/muscle tone, and Respiration. Each sign receives a score between 0 and 2, with high score indicating better health. The Total Apgar Score is calculated by summing the individual aspect scores and ranges from 0 to 10, with higher scores indicating better health.
  score | 8 [7 to 9] | 8 [7 to 9] | 8 [7 to 9]
Number of Infants who Required Oxygen [Count of Participants; unit: Participants]
  No | 71 | 68 | 139
  Unknown | 1 | 1 | 2
  Yes | 344 | 342 | 686
Number of Infants who Required Positive pressure ventilation [Count of Participants; unit: Participants]
  No | 188 | 185 | 373
  Unknown | 0 | 1 | 1
  Yes | 228 | 225 | 453
Number of Infants who Required CPAP [Count of Participants; unit: Participants]
  No | 81 | 81 | 162
  Unknown | 0 | 1 | 1
  Yes | 335 | 329 | 664
Number of Infants who Required Intubation [Count of Participants; unit: Participants]
  No | 370 | 366 | 736
  Yes | 46 | 45 | 91
Number of Infants who Required Chest compressions [Count of Participants; unit: Participants]
  No | 416 | 405 | 821
  Unknown | 0 | 1 | 1
  Yes | 0 | 5 | 5
Number of Infants who Required Epinephrine [Count of Participants; unit: Participants]
  No | 416 | 409 | 825
  Yes | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Days Between Randomization and Hospital Discharge
Description: The number of days between randomization and hospital discharge. This outcome is censored at 48 weeks PMA and at time of transfer or death.
Time Frame: Randomization through hospital discharge, censored at time of transfer, death, or 48 wks PMA
Population: An intent-to-treat (ITT) analysis which included all infants participants who were randomized and who provided outcome data.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Caffeine | Placebo
Number analyzed (Participants) | 415 | 410
days | 18 [10 to 30] | 16.5 [10 to 27]

2. Secondary Outcome: The Number of Days to Physiologic Maturity After Randomization
Description: The number of days to physiologic maturity after randomization. Physiologic maturity is defined: 1. Temperature: out of the incubator for at least 48 hours with normal body temperature; 2. Feeding: oral feeding at a volume of at least 140 ml/kg for 48 hours or growing on less than 140 ml/kg/day for at least 48 hours; 3. Respiratory: apnea-free for at least 5 consecutive days. This outcome is censored at 48 weeks PMA
Time Frame: Randomization through hospital discharge, censored at time of transfer, death, or 48 wks PMA
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Caffeine | Placebo
Number analyzed (Participants) | 390 | 388
days | 13 [7 to 23] | 14 [8 to 23]

3. Secondary Outcome: The Number of Days to When Out of Incubator for 48 Hours: When Maintained Stable Temp for 48 Hrs
Description: The number of days to when out of incubator for 48 hours: when maintained stable temp for 48 hrs. This outcome is censored at 48 weeks PMA
Time Frame: Randomization through hospital discharge, censored at time of transfer, death, or 48 wks PMA
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Caffeine | Placebo
Number analyzed (Participants) | 201 | 199
days | 5 [2 to 9] | 5 [1 to 9]

4. Secondary Outcome: The Number of Days to Apnea/ Bradycardia Free for 5 Consecutive Days
Description: The number of days to apnea/ bradycardia free for 5 consecutive days. This outcome is censored at 48 weeks PMA
Time Frame: Randomization through hospital discharge, censored at time of transfer, death, or 48 wks PMA
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Caffeine | Placebo
Number analyzed (Participants) | 325 | 326
days | 8 [5 to 16] | 11 [5 to 18]

5. Secondary Outcome: The Number of Days to Oral Feeds >140 ml/kg/Day or Growing on Less Than 140 ml/kg/Day for at Least 48 Hours
Description: The number of days oral feeds >140 ml/kg/day or growing on less than 140 ml/kg/day for at least 48 hours. This outcome is censored at 48 weeks PMA
Time Frame: Randomization through hospital discharge, censored at time of transfer, death, or 48 wks PMA
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Caffeine | Placebo
Number analyzed (Participants) | 256 | 251
days | 14 [6 to 23] | 12 [5 to 22]

6. Secondary Outcome: Post-menstrual Age at Discharge
Description: The post-menstrual age of the infant at discharge censored at 48 weeks PMA and at time of transfer or death
Time Frame: Randomization through hospital discharge, censored at time of transfer, death, or 48 wks PMA
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: weeks
Arm/Group | Caffeine | Placebo
Number analyzed (Participants) | 415 | 411
weeks | 37.7 [37.5 to 37.9] | 37.6 [37.4 to 37.8]

7. Secondary Outcome: Weight Gain From Randomization Until Status
Description: Weight gain from randomization until status %(discharge up to 48 wks PMA, with censoring at time of transfer or death%).
Time Frame: Randomization through hospital discharge, censored at time of transfer, death, or 48 wks PMA
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: grams per day
Arm/Group | Caffeine | Placebo
Number analyzed (Participants) | 413 | 410
grams per day | 28.9 [28.1 to 29.8] | 32.2 [30.9 to 33.4]

8. Secondary Outcome: The Number of Days After Randomization Until Status That Infant Had at Least Two Consecutive Heart Rates >200 Documented at Least 3 Hours Apart
Description: The number of days after randomization until status that infant had at least two consecutive heart rates >200 documented at least 3 hours apart
Time Frame: Randomization through hospital discharge, censored at time of transfer, death, or 48 wks PMA
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Caffeine | Placebo
Number analyzed (Participants) | 414 | 411
days | 0 [0 to 0] | 0 [0 to 0]

9. Secondary Outcome: Treatment for High Blood Pressure
Description: Treatment for high blood pressure initiated after randomization until status.
Time Frame: Randomization through hospital discharge, censored at time of transfer, death, or 48 wks PMA
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Caffeine | Placebo
Number analyzed (Participants) | 414 | 411
Participants
  No | 412 | 410
  Yes | 2 | 1

10. Secondary Outcome: The Number of Episodes Between Randomization and Status That Infant Was Placed NPO for >= 24 Hours
Description: The number of episodes between randomization and status that infant was placed NPO for >= 24 hours
Time Frame: Randomization through hospital discharge, censored at time of transfer, death, or 48 wks PMA
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: episodes
Arm/Group | Caffeine | Placebo
Number analyzed (Participants) | 414 | 411
episodes | 0 [0 to 0] | 0 [0 to 0]

11. Secondary Outcome: Use of Anti-reflux Medications
Description: The use of anti-reflux medications started between randomization and status
Time Frame: Randomization through hospital discharge, censored at time of transfer, death, or 48 wks PMA
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Caffeine | Placebo
Number analyzed (Participants) | 414 | 411
Participants
  No | 384 | 387
  Yes | 30 | 24

12. Secondary Outcome: Number of Days That Significant Apnea/Bradycardia
Description: The number of days that significant apnea/bradycardia, as defined by documentation of infant receiving any of the following between randomization and status: open label caffeine, other methylxanthines, doxapram, CPAP or ventilatory support for apnea/bradycardia.
Time Frame: Randomization through hospital discharge, censored at time of transfer, death, or 48 wks PMA
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Caffeine | Placebo
Number analyzed (Participants) | 414 | 410
days | 0 [0 to 0] | 0 [0 to 0]

13. Secondary Outcome: All-cause Mortality
Description: All-cause mortality
Time Frame: Randomization through hospital discharge, censored at time of transfer, death, or 48 wks PMA
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Caffeine | Placebo
Number analyzed (Participants) | 416 | 411
Participants
  No | 415 | 411
  Yes | 1 | 0

14. Secondary Outcome: Number of All-cause Readmissions Within First 4 Weeks Post-discharge
Description: Number of all-cause readmissions within first 4 weeks post-discharge
Time Frame: Discharge through 4 weeks post-discharge
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: count of readmissions
Arm/Group | Caffeine | Placebo
Number analyzed (Participants) | 390 | 397
count of readmissions | 0 [0 to 0] | 0 [0 to 0]

15. Secondary Outcome: Number of All-cause Readmissions Within Second 4 Weeks Post-discharge
Description: Number of all-cause readmissions within second 4 weeks post-discharge
Time Frame: 4 weeks through 8 weeks post-discharge
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: count of readmissions
Arm/Group | Caffeine | Placebo
Number analyzed (Participants) | 390 | 397
count of readmissions | 0 [0 to 0] | 0 [0 to 0]

16. Secondary Outcome: Number of All-cause Readmissions Within First 8 Weeks Post-discharge
Description: Number of all-cause readmissions within first 8 weeks post-discharge
Time Frame: Discharge through 8 weeks post-discharge
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: count of readmissions
Arm/Group | Caffeine | Placebo
Number analyzed (Participants) | 390 | 397
count of readmissions | 0 [0 to 0] | 0 [0 to 0]

17. Secondary Outcome: Number of All-cause Sick Visits, Urgent Care, Emergency Rooms, or Health Care Provider%'s Office, Within First 4 Weeks Post-discharge
Description: Number of all-cause sick visits, urgent care, emergency rooms, or health care provider%'s office, within first 4 weeks post-discharge
Time Frame: Discharge through 4 weeks post-discharge
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: count of sick visits
Arm/Group | Caffeine | Placebo
Number analyzed (Participants) | 390 | 397
count of sick visits | 0 [0 to 0] | 0 [0 to 0]

18. Secondary Outcome: Number of All-cause Sick Visits, Urgent Care, Emergency Rooms, or Health Care Provider%'s Office, Within Second 4 Weeks Post-discharge
Description: Number of all-cause sick visits, urgent care, emergency rooms, or health care provider%'s office, within second 4 weeks post-discharge
Time Frame: 4 weeks through 8 weeks post-discharge
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: count of sick visits
Arm/Group | Caffeine | Placebo
Number analyzed (Participants) | 390 | 397
count of sick visits | 0 [0 to 0] | 0 [0 to 0]

19. Secondary Outcome: Number of All-cause Sick Visits, Urgent Care, Emergency Rooms, or Health Care Provider%'s Office, Within First 8 Weeks Post-discharge
Description: Number of all-cause sick visits, urgent care, emergency rooms, or health care provider%'s office, within first 8 weeks post-discharge
Time Frame: Discharge through 8 weeks post-discharge
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: count of sick visits
Arm/Group | Caffeine | Placebo
Number analyzed (Participants) | 390 | 397
count of sick visits | 0 [0 to 0] | 0 [0 to 0]

20. Primary Outcome: Number of Sick Visits Related to Apneic or Apparent Life-threatening Events Within First 4 Weeks Post-discharge
Description: Number of sick visits related to apneic or apparent life-threatening events within first 4 weeks post-discharge MEASTYPE=SEC
Time Frame: Discharge through 4 weeks post-discharge
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: count of apnea visits
Arm/Group | Caffeine | Placebo
Number analyzed (Participants) | 390 | 397
count of apnea visits | 0 [0 to 0] | 0 [0 to 0]

21. Secondary Outcome: Number of Sick Visits Related to Apneic or Apparent Life-threatening Events Within Second 4 Weeks Post-discharge
Description: Number of sick visits related to apneic or apparent life-threatening events within second 4 weeks post-discharge
Time Frame: 4 weeks through 8 weeks post-discharge
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: count of apnea visits
Arm/Group | Caffeine | Placebo
Number analyzed (Participants) | 390 | 397
count of apnea visits | 0 [0 to 0] | 0 [0 to 0]

22. Secondary Outcome: Number of Sick Visits Related to Apneic or Apparent Life-threatening Events Within First 8 Weeks Post-discharge
Description: Number of sick visits related to apneic or apparent life-threatening events within first 8 weeks post-discharge
Time Frame: Discharge through 8 weeks post-discharge
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: count of apnea visits
Arm/Group | Caffeine | Placebo
Number analyzed (Participants) | 390 | 397
count of apnea visits | 0 [0 to 0] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: Randomization through 8-weeks post discharge, up to 48 weeks Post-Menstrual Age.
Description: Adverse events were collected on all randomized infants from the time of randomization through the end of the post-discharge follow-up (8 weeks post-discharge or 48 weeks post-menstrual age, whichever comes first)
Arm/Group | Caffeine | Placebo
All-Cause Mortality (participants affected / at risk) | 1/416 | 0/411
Serious Adverse Events (participants affected / at risk) | 12/416 | 22/411
Other Adverse Events (participants affected / at risk) | 10/416 | 24/411
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caffeine (N=416) | Placebo (N=411)
Neonatal tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Necrotising enterocolitis neonatal (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (4)
Bronchiolitis (Infections and infestations) | 1 (1) | 2 (2)
Enterovirus infection (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Mastoiditis (Infections and infestations) | 0 (0) | 1 (1)
Meningitis neonatal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia moraxella (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 2 (2) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1) | 2 (2)
Sepsis neonatal (Infections and infestations) | 1 (1) | 2 (2)
Subperiosteal abscess (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection neonatal (Infections and infestations) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Apnea neonatal (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 9 (10)
Cyanosis neonatal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Neonatal hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension neonatal (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caffeine (N=416) | Placebo (N=411)
Arrhythmia neonatal (Cardiac disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Necrotising enterocolitis neonatal (Gastrointestinal disorders) | 0 (0) | 2 (2)
Sepsis neonatal (Infections and infestations) | 0 (0) | 2 (2)
Apnea neonatal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 9 (10)
Hypertension neonatal (Vascular disorders) | 9 (9) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT03340727/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/27/NCT03340727/SAP_002.pdf
  • Informed Consent Form (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT03340727/ICF_003.pdf